CLINICAL TRIAL: NCT06359964
Title: Infective Complications in Transperineal Prostate Biopsy Without Antibiotic Prophylaxis: A Prospective Cohort Study
Brief Title: Infective Complications in TP Biopsy Without Antibiotic Prophylaxis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, CHIU Ka Fung Peter, Associate Professor, Chinese University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRE2023.195
Record Dates: First submitted 2024-03-05; First posted 2024-04-11 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TP BIospy without antibiotic prophylaxis (Experimental): Transperineal Biopsy without antibiotic prophylaxis
  Interventions: Procedure: Transperineal Biopsy without antibiotics prophylaxis
- TP BIospy with antibiotic prophylaxis (Active Comparator): Transperineal Biopsy with antibiotic prophylaxis
  Interventions: Procedure: Transperineal Biopsy with antibiotics prophylaxis

INTERVENTIONS:
Procedure: Transperineal Biopsy without antibiotics prophylaxis — Transperineal Biopsy without antibiotics prophylaxis
  Arms: TP BIospy without antibiotic prophylaxis
Procedure: Transperineal Biopsy with antibiotics prophylaxis — Transperineal Biopsy with antibiotics prophylaxis
  Arms: TP BIospy with antibiotic prophylaxis

SUMMARY:
This study is a prospective cohort study to delineate the infective outcomes and incidence after transperineal prostate biopsy with no antibiotic prophylaxis, compared to the existing data on outcomes on patients receiving transperineal prostate biopsy with antibiotic prophylaxis.

DETAILED DESCRIPTION:
All consecutive patients receiving transperineal prostate biopsy in the PWH will be recruited to the exposure cohort after informed consent. Antibiotic prophylaxis will not be given for patients in the exposure group. All patients will undergo transperineal prostate biopsy in the usual manner and technique, under the Ginsburg protocol. Systematic and MRI-TRUS fusion for systematic plus targeted biopsy will be performed based on the usual clinical indications, depending on the clinical need. Follow-up data will be collected, with particular interest on the assessment of infective complications.

Prospectively collected data will also be retrieved from the electronic patient record (ePR) under the Hospital Authority, to assess relevant information on infective complications for patients who received transperineal prostate biopsy in PWH and NDH from 2019 to 2023. These patients received antibiotic prophylaxis prior to their biopsies, and eligible patients will be included as the control cohort for comparison. Propensity score matching will be utilized in order to create a control group that is similar to the exposure group with balanced baseline. Statistical analysis will be performed on the retrieve data.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients in participating centres receiving transperineal USG-guided biopsy for any indication including:
* Elevated PSA
* Abnormal DRE
* Follow-up biopsy in active surveillance
* Suspicion of CAP recurrence after radiotherapy
* Follow-up biopsy after focal therapy
* Consenting to the study

Exclusion Criteria:

* Recent suspected UTI within 1 month
* Recent culture proven bacteriuria within 1 month
* History of recurrent UTI
* Indwelling urinary catheter
* Immunocompromised state
* High risk of infective endocarditis (including prosthetic heart valve, congenital heart disease, or previous history of infective endocarditis
* Incompetent or incapable of understanding the nature of the study or giving informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 1900 (Estimated)
Dates: Start 2024-08-04 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
The difference in UTI hospitalization rate between the two groups after biopsy | Within 14 days of biopsy
  UTI hospitalization rate is defined symptomology requiring admission to an in-patient facility
The difference in urosepsis rates between the two groups after biopsy | Within 14 days of biopsy
  Urosepsis is defined as sepsis of likely urological source either based on symptomology or bacteriology.

SECONDARY OUTCOMES:
Post-biopsy UTI rates between the two groups | At post-biopsy Day 14
  The result of clean catch mid-stream urine for culture
Assessment of bacteriology and antibiotic resistant profile between the two groups | At post-biopsy Day 14
  The bacteriology and antibiotic resistant profile are assessed by clean-catch urine culture.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Ka-Fung CHIU, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Derin O, Fonseca L, Sanchez-Salas R, Roberts MJ. Infectious complications of prostate biopsy: winning battles but not war. World J Urol. 2020 Nov;38(11):2743-2753. doi: 10.1007/s00345-020-03112-3. Epub 2020 Feb 24. PMID 32095882
- [Background] Li JKM, Wang LL, Lau BSY, Tse RTH, Cheng CKL, Leung SCH, Wong CYP, Tsui SKW, Teoh JYC, Chiu PKF, Ng CF. Oral antibiotics perturbation on gut microbiota after prostate biopsy. Front Cell Infect Microbiol. 2022 Aug 16;12:959903. doi: 10.3389/fcimb.2022.959903. eCollection 2022. PMID 36051239
- [Background] Castellani D, Pirola GM, Law YXT, Gubbiotti M, Giulioni C, Scarcella S, Wroclawski ML, Chan E, Chiu PK, Teoh JY, Gauhar V, Rubilotta E. Infection Rate after Transperineal Prostate Biopsy with and without Prophylactic Antibiotics: Results from a Systematic Review and Meta-Analysis of Comparative Studies. J Urol. 2022 Jan;207(1):25-34. doi: 10.1097/JU.0000000000002251. Epub 2021 Sep 24. PMID 34555932
- [Background] Basourakos SP, Alshak MN, Lewicki PJ, Cheng E, Tzeng M, DeRosa AP, Allaway MJ, Ross AE, Schaeffer EM, Patel HD, Hu JC, Gorin MA. Role of Prophylactic Antibiotics in Transperineal Prostate Biopsy: A Systematic Review and Meta-analysis. Eur Urol Open Sci. 2022 Jan 29;37:53-63. doi: 10.1016/j.euros.2022.01.001. eCollection 2022 Mar. PMID 35243391
- [Background] Jacewicz M, Gunzel K, Rud E, Sandbaek G, Magheli A, Busch J, Hinz S, Baco E. Antibiotic prophylaxis versus no antibiotic prophylaxis in transperineal prostate biopsies (NORAPP): a randomised, open-label, non-inferiority trial. Lancet Infect Dis. 2022 Oct;22(10):1465-1471. doi: 10.1016/S1473-3099(22)00373-5. Epub 2022 Jul 12. PMID 35839791
- [Background] Singhal U, Qi J, Daignault-Newton S, George AK. Antibiotic prophylaxis for transperineal prostate biopsy? An unanswered question. Lancet Infect Dis. 2022 Dec;22(12):1662. doi: 10.1016/S1473-3099(22)00738-1. Epub 2022 Nov 7. No abstract available. PMID 36356605
- [Background] Rassen JA, Shelat AA, Myers J, Glynn RJ, Rothman KJ, Schneeweiss S. One-to-many propensity score matching in cohort studies. Pharmacoepidemiol Drug Saf. 2012 May;21 Suppl 2:69-80. doi: 10.1002/pds.3263. PMID 22552982
- [Background] Kotel'nikov VP. [Current value of the deontologic principles of N. I. Pirogova]. Klin Med (Mosk). 1985 Nov;63(11):131-8. No abstract available. Russian. PMID 3910956
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338